CLINICAL TRIAL: NCT01819805
Title: Evaluation of the Improvement of Pain and Health-Related Quality of Life in Patients With Chronic Non-Malignant Pain Taking Tramadol HCl (75mg)/Acetaminophen (650mg) Extended Release Tablet: Multicenter, Open Label, Prospective, Observational Study
Brief Title: A Study to Assess the Improvement of Pain and Health-Related Quality of Life in Patients With Chronic Non-Malignant Pain Taking Tramadol Hydrochloride and Acetaminophen
Status: Completed | Type: Observational
Sponsor: Janssen Korea, Ltd., Korea (Industry)
Responsible Party: Sponsor
Other Study IDs: CR100722; TRAMAPPAI4047 (Other: Janssen Korea, Ltd., Korea); ULTER-KOR-5005 (Other: Janssen Korea, Ltd., Korea)
Record Dates: First submitted 2013-02-07; First posted 2013-03-28 (Estimated); Last update posted 2015-01-01 (Estimated); Status verified 2014-12

CONDITIONS: Chronic Pain
Keywords: Chronic pain; Chronic non-malignant pain; Non-malignant; Pain; Extended release tablet; Tramadol hydrochloride; Tramadol HCl; Acetaminophen; Ultracet ER
MeSH Terms: conditions — Chronic Pain; Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients taking tramadol hydrochloride and acetaminophen
  Interventions: Drug: No intervention

INTERVENTIONS:
Drug: No intervention — This is an observational study. Patients taking extended release tramadol hydrochloride 75 mg and acetaminophen 650 mg orally twice daily will be observed.
  Other Names: ULTRACET ER

SUMMARY:
The purpose of this study is to evaluate the impact of extended release tramadol hydrochloride (75 mg) and acetaminophen (650 mg) tablets on improvement of pain.

DETAILED DESCRIPTION:
This is a multi-center (study conducted at multiple sites), open label (all people know the identity of the intervention), prospective (in which the participants are first identified and then followed forward as time passes), observational study to assess the improvement of pain and health-related quality of life in patients with moderate to severe chronic non-malignant pain. The study will enroll patients who had already filled a prescription for extended release tramadol hydrochloride 75 mg and acetaminophen 650 mg (ULTRACET ER). The study medication will be administered according to local label insert. The study medication will be taken twice daily, 1 to 2 tablets each time, for a maximum of 4 tablets. Safety evaluations for adverse events will be performed throughout the study. The total duration of the study will be approximately of 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients with the prescription of ULTRACET ER for the treatment of moderate to severe pain
* Complaining of chronic pain for more than 3 months

Exclusion Criteria:

* Patient who had been treated with extended release tramadol hydrochloride (75mg) and acetaminophen (650mg) or strong opioids (eg, morphine, fentanyl, oxycodone, hydromorphone) within the past 4 weeks
* Patient with a severe mental disease and with a medical history of hypersensitivity to opioid analgesics
* Pregnant females or the females likely to become pregnant during the study period
* Patient who had been believed likely to complain of more pain than the real pain he or she is experiencing because of industrial disaster, car insurance, and others
* Patients who are contraindicated according to the warnings, precautions and prohibitions regarding extended release tramadol hydrochloride (75mg) and acetaminophen (650mg)

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic non-malignant pain taking tramadol hydrochloride and acetaminophen
Sampling Method: Non-Probability Sample
Enrollment: 1065 (Actual)
Dates: Start 2011-09; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Number of patients with more than 30 percentage reduction in percentage Pain Intensity Difference (PID) from baseline | Baseline (Week 1) to Week 12
  Numerical Rating Scale (NRS) is an 11-point scale to measure the pain intensity and is used by patients to rate their pain from 0 (absence of pain) to 10 (extreme pain). Percentage PID =[(NRS score at baseline - NRS score at Week 12)/NRS score at baseline] X 100.

SECONDARY OUTCOMES:
Change in scores of Korean version of the EuroQol 5 Dimensional (KEQ-5D) Questionnaire from baseline | Baseline to Week 12
  The KEQ-5D is a validated generic measure of quality of life which usually requires less than 1 minute to complete (eg, the questionnaire may have questions about mobility, self care, usual activities, pain/discomfort and anxiety/depression).
The degree of night sleep disturbance due to pain | Baseline to Week 12
  Sleep disturbance due to pain will be measured using a Numeric Rating Scale (NRS): 1 = None, 10 = Complete.
The degree of Interference with activity of daily living due to Pain | Baseline to Week 12
  The degree of interference with activity of daily living due to pain will be assessed on a 5-point scale: 1 = No interference, 5 = Great interference. Activity of daily living means household work performance, etc.
The degree of Interference with social activities due to Pain | Baseline to Week 12
  The degree of interference with social life performance due to pain will be measured on a 5-point scale; 1 = No interference, 5 = Great interference. Social activities means interpersonal relationship, going out, working life, etc.
The investigator's global assessment of pain treatment | Week 4 to Week 12
  The investigator will assess on a 5-point scale (1= not effective, 5= greatly effective) how effective the study drug has been for a patient, in the judgment of the investigator.
The patient's global assessment of pain treatment | Week 4 to Week 12
  The patient will assess on a 5-point scale (1= not effective, 5= greatly effective) how effective the study drug has been in the judgment of the study patient.
The number of patients who experience adverse events as a measure of safety and tolerability | Week 4 to Week 12

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Korea, Ltd., Korea Clinical trial, Study Director — Janssen Korea, Ltd., Korea
Locations (14):
- South Korea (14):
  - Busan
  - Cheonan
  - Chungcheongbuk-Do
  - Chungju
  - Daegu
  - Daejeon
  - Goyang
  - Gyeonggi-do
  - Hwasun Gun
  - Kwangiu
  - Kwangjoo
  - Kyungjoo
  - Seoul
  - Suwon